CLINICAL TRIAL: NCT00478582
Title: Validation of a New Standardized Clinical Anemia Evaluation Score Using a Hb Visual Scale in Nephrological Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: HB 5/2007
Record Dates: First submitted 2007-05-24; First posted 2007-05-25 (Estimated); Last update posted 2011-01-13 (Estimated); Status verified 2011-01

CONDITIONS: Anemia
Keywords: Anemia; Visual scale; nephrological patients; Anemia in nephrological patients
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Estimation of Hb concentrations with the HemoHue card

SUMMARY:
The clinical evaluation of anemia is usually done by examination of the palpebral conjontivae coloration. This appreciation remains crude and largely observer dependent, as no reference scale was successfully proposed,. A Hb visual scale allowing the assessment of the degree of clinical anemia has been developed. Its use has been validated so far in small patient groups in the following settings: blood donation, cardiac surgery, oncology and consultation of general practitioners.

The objective of the present investigation is to validate the use of a Hb visual scale for the clinical evaluation of anemia in patients with kidney disease patients

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronich kidney disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-05; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Comparison of visual estimated Hb concentrations with measured Hb concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Dominik Uehlinger, Prof, Study Director; Dominik Uelinger, Prof, Principal Investigator
Locations (1):
- Department of nephrology and hypertension, University hospital of berne, Bern, Canton of Bern, Switzerland